CLINICAL TRIAL: NCT04098419
Title: Evaluation of a Two-tiered Cross-age Teaching Model for Food Literacy-based Education
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Discontinuing the study because of COVID-19
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1473718
Record Dates: First submitted 2019-09-09; First posted 2019-09-23 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Food Literacy; Adolescent Health; Cross-age Teaching; Nutrition Education; Experiential Learning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Williams Implementation (Experimental)
  Interventions: Behavioral: Science for Life
- Pittsburg Implementation (Experimental)
  Interventions: Behavioral: Science for Life

INTERVENTIONS:
Behavioral: Science for Life — The implementation for both school years will follow the same procedures with different cohorts. Sixteen adolescents will be recruited through existing after-school programs at each location (32 total each year). College interns will facilitate food literacy lessons after school once per week with high school-aged adolescents. Beginning in January, adolescents will participate in training led by project staff and college interns to become competent cross-age teachers for garden-enhanced nutrition curricula. This training will consist of instruction in utilization of inquiry-based teaching practices and will be followed by adolescents practicing facilitating the curricula in teaching pairs. Up to 32 younger youth participants at each location (up to 64 total each year) will be recruited from local elementary schools while adolescents complete the cross-age teaching training. With mentorship from college interns, adolescents will facilitate curricula in pairs with younger youth.

SUMMARY:
This project will serve adolescents from low-income and historically underserved communities through expansion of existing after-school programs. Adolescents from these communities tend to have slower academic progression and higher high school dropout rates. Extracurricular activities, including informal education through after-school programming, have been suggested to improve these rates and increase college enrollment by supporting traditional classroom-based education. The proposed project aims to educate high school-aged adolescents in food, agriculture, natural resources, and human (FANH) sciences through informal food literacy education. The project also includes a two-tiered cross-age teaching model, allowing for adolescents to be educated by college interns and to become educators for younger youth. Existing curricula, that encompass FANH sciences, will be utilized at each stage of the project. The purpose of the project is not only to educate adolescents in FANH sciences, but also to advance their motivation and efficacy for graduating high school, attending college, and majoring in FANH sciences. The project aims to accomplish these objectives through empowering adolescents to obtain knowledge, skills, and excitement for food literacy. As this model has not been utilized previously, this project will produce a best practices guide for implementing the existing curricula within a two-tiered cross-age teaching model. Additionally, the college internship and mentoring program created through this project will be continued at the initial sites and expanded to other communities. This will allow for a sustainable approach to educating adolescents in FANH sciences and providing mentorship that encourages future enrollment in college.

ELIGIBILITY:
Inclusion Criteria:

* There are two groups of participants (adolescents and younger youth) that will be recruited for this study. Adolescent participants must be high school-aged, approximately 13-17 years. Younger youth must be upper elementary school-aged, approximately 9-12 years. Participants for both age groups will be recruited from existing afterschool programs within each participating school district. Comparison youth for both age groups will be recruited from other students within the same school districts.

For the 2019-2020 and 2020-2021 school years, the participating school districts will be in Pittsburg and Williams, California.

Exclusion Criteria:

* Youth from other school districts

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Nutrition Knowledge | 1 school year
  Assessed using age-specific validated questionnaires. The score on this assessment is presented as a percentage of correct responses out of 30 questions. Higher percentages represent a better outcome.
Self-Efficacy about Teaching Nutrition | 5 months
  Adapted questionnaire to assess teen self-efficacy about teaching nutrition using a retrospective, post-then-pre method. This assessment features a 5-point Likert scale.
Self-Efficacy about Cooking Skills | 1 school year
  Motivation and cooking confidence will be measured using an adapted version of a questionnaire developed by University of Louisiana. This questionnaire assesses intrinsic motivation to cook and perceived competence using a retrospective, post-then-pre method.This assessment features a 5-point Likert scale.
Fruit and Vegetable Intake (Skin Carotenoids) | 1 year
  Fruit and vegetable consumption will be collected using reflection spectroscopy through an instrument called "Veggie Meter." The Veggie Meter can be utilized to objectively estimate carotenoid-containing fruit and vegetable consumption through measurement of skin carotenoids in the fingertip. A handout about this tool will be provided to parents/guardians with the consent form. For the most reliable results, this measurement will be collected during the same time of year to limit false results due to seasonal changes in dietary pattern.
Dietary intake | 1 school year
  A commonly used food frequency questionnaire will be utilized to measure dietary intake in adolescents and younger youth (Block Kids 2004). The tool has been determined to be appropriate for ages 7-17 years. To best assess the eating pattern of the target populations, the option for inclusion of food commonly eaten by Hispanic populations has been selected. This assessment tool will be provided in both English and Spanish so that parents/guardians can help participants complete the assessment at home. Additionally, serving size references will be sent home with the questionnaire. This assessment includes a variety of foods and asks participants how many days in the last week they consumed each food.

SECONDARY OUTCOMES:
Household Food Security | 1 school year
  Household food security will be measured using the USDA's U.S. Household Food Security Survey Module. This widely utilized 12-item module has been modified to a fillable questionnaire for parents or guardians of youth to complete.
Anthropometrics (to calculate BMI) | 1 school year
  Height, and weight will be measured and used to calculate BMI percentile and BMI-z scores. Participants will be measured in light outdoor clothing after the removal of shoes. Height will be measured to the nearest 0.1cm using a transportable stadiometer and body weight will be measured to the nearest 0.1kg using an electronic scale. Waist circumference will be measured to the nearest cm using a body circumference measuring tape. Adiposity and obesity risk will be assessed via age- and sex-specific BMI percentile as recommended by the Expert Committee on Childhood and Adolescent Overweight and Obesity.
Civic Responsibility | 1 school year
  Civic responsibility will be measured using a reliable questionnaire developed as a part of the 4-H Youth Development Program Healthy Living Measures by the Service-Learning Research and Development Center at University of California, Berkeley. The 24-item questionnaire assesses civic responsibility by measuring three key aspects: connection to community, civic awareness, and civic efficacy. This assessment features a 6-point Likert scale.
Motivation for Educational Attainment | 1 school year
  Motivation and self-efficacy for attaining higher education will be measured using the Adolescent Education Aspirations Questionnaire. This 16-item questionnaire assesses adolescents' motivation and self-efficacy to graduate high school and attend college. This assessment features a 5-point Likert scale.
Academic self-efficacy | 1 school year
  The Academic Self-Efficacy Scale was developed based on the Social Cognitive Theory and found reliable when tested in Indian adolescents. The instrument also demonstrated face and content validity. While translated to English, the tool needed further revision to be appropriate for American adolescents.
Social and emotional self-efficacy | 1 school year
  Portions of the Self-Efficacy Questionnaire for Children (SEQ-C) will be utilized to assess social and emotional self-efficacy. While originally developed in the Netherlands, this questionnaire was tested in two large samples of American adolescents in middle school and high school and found to be an appropriate tool with minor revisions. With assessment of academic self-efficacy being completed with the previously mentioned questionnaire, items referring to academics have been removed from this tool.
Disposition toward FANH sciences | 1 school year
  Disposition toward FANH sciences will be assessed using a modified version of the STEM Semantics Survey. This five-part survey has been shown to reliably measure disposition toward STEM in high school-aged adolescents.
Self-esteem and locus of control | 1 school year
  Self-esteem will be assessed in the high school-aged adolescents and perceptions of locus of control will be measured in both adolescents and younger youth using previously used tools.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Davis, California, United States